CLINICAL TRIAL: NCT01761773
Title: A Phase 1, Open-Label, Parallel-Cohort, Single-Dose Study to Assess the Pharmacokinetics of Cabozantinib (XL184) Capsules in Subjects With Impaired Renal Function
Brief Title: A Single-Dose Study to Assess the Pharmacokinetics of Cabozantinib (XL184) Capsules in Subjects With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL184-017
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Healthy; Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): Subjects with normal renal function: healthy normal adult subjects with an eGFR ≥ 90 mL/min/1.73m2.
  Interventions: Drug: cabozantinib
- Group 2 (Experimental): Subjects with mild renal impairment: adult subjects with a eCFR ≥ 90 mL/min/1.73m2.
  Interventions: Drug: cabozantinib
- Group 3 (Experimental): Moderate renal impairment: adult subjects with an eGFR between ≥30 - ≤ 59 mL/min/1.73m2.
  Interventions: Drug: cabozantinib
- Group 4 (Experimental): Severe renal impairment: adult subjects with an eGFR ≤ 29 mL/min/1.73m2, not on dialysis.
  Interventions: Drug: cabozantinib

INTERVENTIONS:
Drug: cabozantinib — 3 20-mg strength capsules (60 mg dose) administered as a single oral dose on Day 1 of study participation.
  Other Names: XL184

SUMMARY:
The main objective of the trial is to compare the pharmacokinetics of a 60 mg dose of cabozantinib in adult subjects with impaired renal function compared with healthy adult subjects. Another objective is to assess the safety and tolerability of cabozantinib in these adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight must be ≥ 50 kg and < 130 kg with a BMI ≤ 38.0 (kg/m2).
* Must use acceptable form of birth control during the course of the study and for 3 months following the single dose of study drug.
* Female subjects of childbearing potential must have a negative pregnancy test at screening and check-in.
* Negative test for HIV; hepatitis A, B, and C.
* Must have adequate vital sign reads at screening and check-in.
* Must be able to comply with dietary and fluid restrictions required for the study.

Exclusion Criteria:

* History of medical or surgical conditions that would interfere with GI absorption, distribution, metabolism, or excretion of the study drug.
* Recent clinical evidence of pancreatic injury.
* Recent use of drugs known to significantly inhibit or induce P450 CYP3A4 enzymes.
* Previous diagnosis of malignancy.
* Unwilling to forgo use of any over-the-counter or non-prescription preparations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Days 1 - 8 as well as the morning of Days 11, 13, 15, 18, 21, 22.
  AUC, Cmax, tmax, kel, t1/2, CL/F, V/F and fu as measure of a single oral 60 mg dose of cabozantinib in adults with impaired renal function compared with healthy subjects matched for age, gender, and body mass index (BMI).
  Subjects will receive a single oral 60 mg dose of cabozantinib on Day 1 and then undergo periodic assessments Days 1 - 8 following this single dose, as well as on the mornings of Days 11, 13, 15, 18, 21, 22.

SECONDARY OUTCOMES:
Safety and Tolerability | Days 1 - 8 and Days 11, 13, 15, 18, 21, 22.
  Number of participants with adverse events, serious adverse events, and laboratory abnormalities as a measure of the safety and tolerability of a single oral 60 mg dose in adult subjects with impaired renal function and in healthy adult subjects.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Miami, Florida
  - Orlando, Florida
  - Neptune City, New Jersey